CLINICAL TRIAL: NCT06024473
Title: A rTMS and Virtual Reality Based Cognitive Rehabilitation Program for MCI
Acronym: rTMS+iVCT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Central Arkansas Veterans Healthcare System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1762307
Record Dates: First submitted 2023-08-24; First posted 2023-09-06 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Mild Cognitive Impairment; Caregiver Burden; Mental Health Issue; ADL; Quality of Life
Keywords: repetitive Transcranial Magnetic Stimulation; immersive virtual reality; Neuropsychiatric Symptoms; Mild Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction; Caregiver Burden

STUDY DESIGN:
Intervention Model Description: 10 participants each will be assigned to the standard treatment, rTMS only or rTMS and iVCT groups
Masking Description: This is an open label pilot study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Standard Treatment (No Intervention): This arm will be followed without intervention
- rTMS (Active Comparator): This group will be randomized to receive rTMS treatment
  Interventions: Device: rTMS
- rTMS+iVCT (Experimental): This group will be randomized to receive rTMS and iVCT treatment
  Interventions: Device: rTMS+iVCT

INTERVENTIONS:
Device: rTMS — Transcranial Magnetic Stimulation
  Arms: rTMS
Device: rTMS+iVCT — Transcranial Magnetic Stimulation and immersive virtual reality
  Arms: rTMS+iVCT

SUMMARY:
This clinical trial is being conducted to see if brain stimulation and brain training together improves cognitive functioning and mood in older adults diagnosed with Mild Cognitive Impairment (MCI). Brain stimulation will be done using repetitive Transcranial Magnetic Stimulation (rTMS). Brain training will be done using immersive virtual reality cognitive training (iVCT) program. The goals of this clinical trail are as follows:

* Examine if rTMS+iVCT intervention can improve and sustain objective cognitive functioning in individuals with MCI more than control or rTMS only groups
* Examine if rTMS+iVCT intervention improves participants mental health symptoms, functional abilities, and quality of life more than control or rTMS only groups
* Examine the impact of rTMS+iVCT intervention on caregiver burden.

Eligible participants will be assigned to a standard treatment (no intervention control) group, rTMS only group of rTMS+iVCT group. All participants will undergo baseline assessment to evaluate their cognitive, emotional, and functional abilities. Those in the rTMS only group will receive rTMS treatments for five days per week for two weeks (total of ten sessions). Those in the rTMS+iVCT group will receive rTMS treatment followed by iVCT training for five days a week for two weeks (total of ten sessions). All participants will then repeat testing 2 weeks and three months after baseline testing to assess for possible treatment related changes and lasting effects.

DETAILED DESCRIPTION:
The primary objective of this pilot study is to assess if combined treatment with repetitive transcranial magnetic stimulation (rTMS) and immersive virtual reality mediated cognitive training program (iVCT) improves cognitive, emotional, and functional abilities in participants with mild cognitive impairment (MCI) compared to usual care. Secondary objective of the study is assess if rTMS+iVCT treatment improves caregiver burden.

Older Veterans (N=50) age ≥ 55 years with mild cognitive impairment will be recruited. All participants will be screened for suitability for the rTMS and iVCT treatments. Those eligible (N=30) will complete a baseline assessment of their cognitive, emotional, and functional abilities and caregiver burden (Visit 1). Participants (N=30) will be randomly assigned to a rTMS group, rTMS+iVCT group, and control group.. Participants in the rTMS group will receive rTMS treatment daily for 5 days of the week for 2 weeks. Participants in the rTMS+iVCT group will receive rTMS treatment followed by 30-60 minutes of iVCT intervention daily for 5 days of the week for 2 weeks. Participants in the control group will receive usual care. All testing will be repeated posttreatment at 2 weeks (Visit 2) and at 3 months(Visit 3) .

Innovations include combination of two non-pharmacological interventions and the inclusion of 3-month post-treatment testing to assess the durability of changes. Feedback will be gathered to improve the treatment program. Assuming positive findings, this research will help establish a new treatment modality for improving the cognitive, emotional, and functional abilities in MCI.

ELIGIBILITY:
Inclusion Criteria:

* age 55 and over
* previous diagnosis of Mild Cognitive Impairment
* Score of 18 or over on the MoCA during pre-screening procedures.

Exclusion Criteria:

* below 55 years old
* Do not pass the TMS Adult Safety Screening
* Taking medications known to increase risk of seizure
* Taking ototoxic medications
* Those with implanted device
* History of bipolar disorder
* History of Tourette's syndrome or presence of motor tics
* History of seizures/ seizures in first degree relatives
* History of stroke, aneurysm, or cranial neurosurgery
* Current alcohol related disorder needing medical treatment
* History of abnormal electroencephalogram (EEG)
* History of motion sickness, nausea, vomiting, seizures, or migraine
* Significant balance/gait impairments/history of falls
* History of hyperacusis or photophobia

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-03-31 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Change in Hopkins Verbal Leaning Test Standard Score | baseline, 2 weeks, 3 months
  range: <55 to >130 - higher score is improvement

SECONDARY OUTCOMES:
Change in NPI | baseline, 2 weeks, 3 months
  Range: 0-33 Lower score is improvement
Change in Functional Activities Questionnaire score | baseline, 2 weeks, 3 months
  Range: 0-30 Lower score is improvement

CONTACTS AND LOCATIONS:
Locations (1):
- Central Arkansas VA Healthcare system, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No
To ensure participant confidentiality, the database will not be made available for public access. One year post completion of the funded study or upon acceptance of the data for publication, deidentified data will be made available to interested parties. Raw data from neuropsychological testing will only be provided to qualified researchers (e.g. neuropsychologists) to prevent misrepresentation. All other data gathered related to clinical, medical, mental health, and psychosocial histories (sans confidential identifiers) will be made available by the PI or research mentor for future research. The PI and research mentor will assume responsibility for ensuring that participant confidentiality is maintained. Prior to release of data, investigators will need to consent to a VA supported data sharing agreement.